CLINICAL TRIAL: NCT01756820
Title: Single-portal Endoscopic Carpal Tunnel Release vs Knifelight for Carpal Tunnel Syndrome. A Randomized Control Trial.
Brief Title: Single-portal Endoscopic Carpal Tunnel Release Versus Knifelight for Carpal Tunnel Syndrome. A Randomized Control Trial
Acronym: CTS-HV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The principal investigator of the study relocated to another institution.
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Haris S Vasiliadis, MD, PhD, Lecturer in Orthopaedics, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ioannina-CTS-HV
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; transverse ligament; carpal tunnel release; endoscopic; minimal invasive; mini-open; median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-portal Endoscopic Carpal Tunnel Release (Microaire®) (Active Comparator): Single-portal Endoscopic Carpal Tunnel Release (Microaire®) will be used, according to the endoscopic technique described by Agee at al.
  Interventions: Procedure: Single-portal Endoscopic Carpal Tunnel Release (Microaire®)
- Knifelight® (Active Comparator): A mini-open technique will be performed, using the Knifelight® (Stryker).
  Interventions: Procedure: Knifelight

INTERVENTIONS:
Procedure: Single-portal Endoscopic Carpal Tunnel Release (Microaire®) — SmartRelease® ECTR endoscopic carpal tunnel release system of MicroAire (http://www.microaire.com/products/ectr-endoscopic-carpal-tunnel/smart-release-ctrs/).
  Other Names: SmartRelease® ECTR endoscopic carpal tunnel release system of MicroAire.
  Arms: Single-portal Endoscopic Carpal Tunnel Release (Microaire®)
Procedure: Knifelight — A mini-open single portal technique using the Knifelight® device (Stryker) according to the surgical technique as described by the manufacturer (antegrade approach)
  Other Names: Knifelight®, Stryker
  Arms: Knifelight®

SUMMARY:
The purpose of this study is to determine whether Single-portal Endoscopic Carpal Tunnel Release (Agee technique, SmartRelease™, MicroAire) and mini-open technique (Knifelight®, Stryker) are equally effective and safe surgical options for the treatment of primary Carpal Tunnel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* primary Carpal Tunnel Syndrome
* no symptoms' relief after 3 months of conservative treatment (NSAIDS, Cast, rest)

  * electrophysiological examination confirms the Carpal Tunnel Syndrome

Exclusion Criteria:

* Secondary Carpal Tunnel Syndrome
* Pregnancy
* Rheumatoid diseases
* Previous trauma at hand or other condition that may effect the anatomy (eg infections)

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Overall Satisfaction | at 1 and 6 months postoperatively
  Satisfaction will be assessed by two ways
  * by answering to the question "are you happy with the result of the surgery?"
  * with a VAS score (0-100) assessing the satisfaction
Complications | up to 6 months postoperatively
  Any complication will be reported including remaining numbness, pain in incision, painful scar, complex regional pain syndrome, infection etc

SECONDARY OUTCOMES:
Pain | at 1 and 6 months postoperatively
  Pain will be assessed
  * as a dichotomous outcome (yes/no)
  * as a continuous outcome (VAS score)
Grip strength | at 1 and 6 months postoperatively
key pinch | at 1 and 6 months postoperatively
Time to return to Activities of Daily Living (ADL) and return to work | up to the end of the study
  Time to return to Activities of Daily Living (ADL) will be reported. Return to work will also be reported for participants that are employed.
Recurrences and reoperations | up to the end of study
Symptom Severity Scale (SSS) | at 1 and 6 months postoperatively
Function Severity Status (FSS) | at 1 and 6 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Haris S Vasiliadis, MD, PhD, Principal Investigator — Department of Orthopaedics, School of Medicine, University of Ioannina, Greece; Theodoros Xenakis, Study Chair — Department of Orthopaedics, School of Medicine, University of Ioannina, Greece; Grigorios Mitsionis, Study Director — Department of Orthopaedics, School of Medicine, University of Ioannina, Greece
Locations (1):
- University Hospital of Ioannina, Ioannina, Greece